CLINICAL TRIAL: NCT05297071
Title: Longitudinal Monitoring of Microsurgical Socket Augmentation Healing With Ultrasonography - A Randomized Controlled Trial
Brief Title: Longitudinal Monitoring of Microsurgical Socket Augmentation Healing With Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Delta Dental Foundation (Other)
Responsible Party: Principal Investigator, Hsun-Liang Chan, Assistant Program Director, Periodontics Graduate Program, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00195615
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Healing Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental Loupes (Other): The surgeon will use dental loupes with a head lamp during the subject's tooth extraction and socket grafting.
  Interventions: Device: Orascopic HDL 3.0 Loupes
- Surgical microscope (Other): The surgeon will use a surgical microscope (with built-in lighting) during the subject's tooth extraction and socket grafting.
  Interventions: Device: Semorr DOM3000D Operation Microscope

INTERVENTIONS:
Device: Orascopic HDL 3.0 Loupes — The loupes will be used during the surgical procedure on half of the subjects. The other half will be performed with a microscope.
  Arms: Dental Loupes
Device: Semorr DOM3000D Operation Microscope — The microscope will be used during the surgical procedure on half of the subjects. The other half will be performed with loupes.
  Arms: Surgical microscope

SUMMARY:
The purpose of this study is to assess healing after tooth extraction with simultaneous socket augmentation (bone grafting during the same appointment as the extraction) when the surgeon uses a surgical microscope, compared to when the surgeon uses dental loupes (magnifiers that are mounted on the surgeon's glasses). These devices magnify and shine light on the area where the surgeon operates.

DETAILED DESCRIPTION:
After a tooth is extracted, a hole is left in the bone called a socket. During the first year of healing after a tooth extraction, there may be up to 60% loss of bone volume at the site. Loss of bone at the edentulous ridge (toothless area) may make it more difficult to place dental implants later. Dental socket grafting is performed to reduce bone resorption after tooth extraction. Grafting involves filling the socket with bone graft (donated human cadaver derived) and covering it with a protective collagen membrane. This graft prevents resorption of the ridge and is slowly replaced with the patient's own bone. The investigators will be trying to determine if bone healing is better if the surgeon uses more powerful magnification.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Single maxillary or mandibular hopeless tooth (a maxillary or mandibular anterior tooth or premolar) planned for extraction due to periapical pathology with a minimum ≥2 mm of the size of the periapical radiolucency shown on a peri-apical film.
3. The patient is planned for implant restoration for the hopeless tooth
4. The study site allows for implant placement with or without additional bone augmentation procedures after the healing
5. Adequate edentulous space for the final restoration on the implant

Exclusion Criteria:

1. Current smokers or quit smoking less than 6 months
2. Major or uncontrolled medical conditions, e.g. poorly controlled diabetes mellitus (HbA1c >8.0%, uncontrolled systemic disease or condition known to alter bone metabolism, e.g. osteoporosis, osteopenia, hyperparathyroidism, Paget's disease, etc.
3. Pregnancy, breast-feeding, could be pregnant or planning to become pregnant in the next 4 months (self-reported)
4. Taking medications known to modify bone metabolism (i.e. bisphosphonates, corticosteroids, hormone replacement therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Bone quality | 12 weeks
  Difference in bone density from the CBCT and ultrasound

SECONDARY OUTCOMES:
Patient-reported outcomes | 1 week, 2 weeks, and 4 weeks
  Difference in patient-reported outcomes. Subjects will be given a questionnaire to evaluate pain perception, pain medication use, and complications after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hsun-Liang Chan, DDS, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States